CLINICAL TRIAL: NCT06054620
Title: The Effect of Exercise and Presleep Nutrition on Muscle Connective Tissue Remodelling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CVC
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Interventional
Keywords: Collagen; Vitamin C; Carbohydrate placebo
MeSH Terms: interventions — Collagen; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Crossover to receive Collagen and Vitamin C (CVC) or Carbohydrate placebo. Unilateral leg exercise (EX) to give 4 outcomes. (1) CVC-EX; (2) CVC-REST; (3) PLACEBO-EX; (4) PLACEBO-REST
Masking Description: Double blinded (investigators and participants). A lab member external to the investigation will code items for the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen and Vitamin C (Active Comparator)
  Interventions: Dietary Supplement: Collagen and Vitamin C
- Carbohydrate Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Carbohydrate Placebo

INTERVENTIONS:
Dietary Supplement: Collagen and Vitamin C — Collagen-modelled crystalline amino acids (30g total, 8g glycine) and vitamin C (500 mg).
  Other Names: CVC
  Arms: Collagen and Vitamin C
Dietary Supplement: Carbohydrate Placebo — Iso-caloric Placebo (30g maltodextrin).
  Arms: Carbohydrate Placebo

SUMMARY:
The primary objective of this study will be to determine the influence of a presleep vitamin C-enriched, collagen-modelled supplement (CVC) on the metabolic fate of dietary glycine using a [2H5]glycine tracer within the intramuscular connective tissue at rest and after a bout of resistance exercise. Other outcomes will be related to regulation collagen remodelling in skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, recreationally active, male and female participants.
* Healthy will be defined as someone who does not have a health condition that would compromise their ability to safely participate in the strenuous physical activity involved in our study as screened for by the Get Active Questionnaire.
* Willing to abstain from resistance exercise for 2 weeks prior to the first metabolic trial and for the duration of the study.
* Participants must be able to abstain from lower-body resistance and/or plyometric exercise for at least 2 weeks prior to the first metabolic trial.
* Participants will be aged 18-35 years old.
* Participants must be normal to overweight (e.g., BMI 18.5-30).
* Participants are willing to abide by the compliance rules of this study (e.g., abstain from physical activity and alcohol 48h prior to each trial).
* Self-reported regular menstrual cycle (25-35d) within the last 3 months (female participants).

Exclusion Criteria:

* Inability to adhere to any of the compliance rules judged by principal investigator or medical doctor.
* Self-reported regular tobacco use.
* Self-reported illicit drug use (e.g. growth hormone, testosterone, etc.).
* Regular use of anti-inflammatory drugs (e.g., ibuprofen).
* Self-reported regularly sleeping less than an average of 7 hours over 3 days (minimum recommended daily amount).
* Individuals who have participated in studies within the past year involving any of the stable isotopes in the study.
* Use of birth control and discontinued use in the last 3-months (female only).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Enrichment of Muscle Collagen | 9 hours
  Overnight incorporation of orally ingested amino acid tracer (D5 Gly and D5 Phe) into mature collagen protein isolated from skeletal muscle biopsy samples taken 9 hours after consumption of the tracer-containing supplement (CVC or PLA) and rest or resistance exercise. Enrichment will be quantified via tandem LC-MS/MS.

SECONDARY OUTCOMES:
Area of muscle with localized collagen remodelling | 9 hours
  Immunofluorescence determined localization of collagen breakdown and synthesis using collagen hybridizing peptide and procollagen antibodies, respectively, on human skeletal muscle cross-sections.
Concentration of Urinary Growth Hormone | 8 hours
  Urine will be collected overnight to measure growth hormone secretion using chemiluminescence.
Enrichment of Myofibrillar Protein | 9 hours
  Overnight incorporation of orally ingested amino acid tracer (D5 Gly and D5 Phe) into myofibrillar proteins isolated from skeletal muscle biopsy samples taken 9 hours after consumption of the tracer-containing supplement (CVC or PLA) and rest or resistance exercise. Enrichment will be quantified via tandem LC-MS/MS.

OTHER OUTCOMES:
Intensity of Muscle Soreness | 24 hours
  Subjective muscle soreness will be quantified using a visual analog scale on trial day mornings and evenings as well as before and after exercise. Using a line spanning 0 to 100 (100 being greatest soreness), participants will select a spot on the line indicating their subjective muscle soreness.

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No